CLINICAL TRIAL: NCT04040998
Title: Compensatory Cognitive Training for Psychosocial Correlates and Self-stigma in Persons With Schizophrenia
Brief Title: Compensatory Cognitive Training For Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Responsible Party: Principal Investigator, YU SHIUAN LIAW, Occupational Therapist, Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TaoyuanMH
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; compensatory cognitive training; generalized estimating equation; psychosocial correlates; self-stigma
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCT+TAU group (Experimental): The participants in CCT+TAU group received compensatory cognitive training plus treatment as usual. The CCT intervention consisted of two 50-minute sessions each week for 10 weeks
  Interventions: Behavioral: Compensatory Cognitive Training
- TAU group (No Intervention): The participants in TAU group received usual treatment at the same time as CCT+TAU group.

INTERVENTIONS:
Behavioral: Compensatory Cognitive Training — Teach the participants compensatory cognitive skills and strategies
  Arms: CCT+TAU group

SUMMARY:
This study aimed to investigate the effects of compensatory cognitive training plus treatment as usual (CCT+TAU) versus treatment as usual (TAU) on on self-esteem, self-efficacy, quality of life, and self-stigma for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, based on the ICD-10 diagnostic criteria for research (World Health Organization, 1992)
* age from 20 to 65
* attending day care center regularly for at least 3 months
* taking stable dose of medication for at least 3 months

Exclusion Criteria:

* comorbid autism spectrum disorder
* comorbid mental retardation
* lacking the reading and writing skills

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Rosenberg Self-Esteem Scale (RSES) | 3 times: 1 to 2 weeks before intervention, 1 day after intervention and at 1 month after intervention
  The Chinese version of Rosenberg Self-Esteem Scale (RSES) was implemented as self-esteem measures. The total score ranged from 10 to 40, with higher scores reflecting higher levels of self-esteem.
Change scores of General Self-Efficacy Scale (GSES) | 3 times: 1 to 2 weeks before intervention, 1 day after intervention and at 1 month after intervention
  The Chinese version of General Self-Efficacy Scale (GSES) consisted of 10 items, assessing optimistic self-beliefs to cope with a variety of difficult demands in life. The total score ranged from 10 to 40, with higher scores indicating more self-efficacy.
Change scores of Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) | 3 times: 1 to 2 weeks before intervention, 1 day after intervention and at 1 month after intervention
  The Chinese version of Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) was administered to measure subjective quality of life. The total scores ranged from 33-165, with higher scores indicating comparatively lower quality of life.
Change scores of Internalized Stigma of Mental Illness (ISMIS) | 3 times: 1 to 2 weeks before intervention, 1 day after intervention and at 1 month after intervention
  The Chinese version of Internalized Stigma of Mental Illness (ISMIS) consists of 29 items incorporated in five domains: alienation, stereotype endorsement, discrimination experience, social withdrawal, and stigma resistance. The total scores range from 29-116. The higher scores on the ISMIS indicates more severe internalized stigmatization.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan Psychiatric Center Ministry of Health and Welfare, Taoyuan District, Taiwan